CLINICAL TRIAL: NCT04707183
Title: Comparison of Continuous Intravenous Lidocaine Infusion Versus ESP Block for Rib Fracture Analgesia
Acronym: Rib Fract ESP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Professor of Anesthesiology, Perioperative and Pain Medicine, Stanford University, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 53844
Record Dates: First submitted 2020-12-23; First posted 2021-01-13 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Rib Fractures
MeSH Terms: conditions — Rib Fractures | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Arm (Placebo Comparator): 1.0mg/kg/hr IV lidocaine infusion
  Interventions: Drug: Lidocaine IV Infusion
- Treatment Arm (Experimental): 10 mL of 2% lidocaine via ESPB
  Interventions: Drug: 2% Lidocaine via ESPB

INTERVENTIONS:
Drug: Lidocaine IV Infusion — Lidocaine will infused through erector spinae plane block catheter in patients with traumatic rib fracture.
  Other Names: Lidocaine
  Arms: Control Arm
Drug: 2% Lidocaine via ESPB — 10 ml of 2% lidocaine will be infused through ESPB in treatment group
  Arms: Treatment Arm

SUMMARY:
Recently in 2016, a new interfascial plane nerve block was developed for thoracic analgesia known as the erector spinae plane block (ESPB). Since its development for thoracic neuropathic pain, the ESPB has been shown to be effective in pain control in multiple procedures including thoracotomies. However, there have been a few published case reports of using ESPB for analgesia in rib fracture management and only one retrospective study which demonstrated improved NRS pain scores and increased incentive spirometry volumes (ICV) post-ESPB compared to pre-ESPB values.

The goal of this study is to compare the effectiveness of ESPB as an alternative method to the current standard of care at Stanford Health Care (SHC) for pain management in traumatic rib fractures. At the investigator's institution, the current standard of care is intravenous (IV) and enteral multimodal analgesia that consists primarily of opioids and a continuous IV lidocaine infusion. Although IV lidocaine has shown some benefit in improving post-surgical pain scores, evidence for its use in MRF is lacking. The purpose of this study is to perform a randomized clinical trial comparing outcomes in pain control and incentive spirometry volumes between continuous ESPB catheters and IV lidocaine infusions in adult patients with acute traumatic rib fractures.

The investigators want to determine if ESPB can provide improved pain control in patients admitted for traumatic rib fractures compared to IV Lidocaine. The aim is to evaluate the clinical effectiveness of ESPB on OME consumption, pain scores, incentive spirometry volumes, cough strength, respiratory complications, inflammatory biomarkers and hospital LOS. Findings from this study can help improve analgesia, quality of care, and patient satisfaction at Stanford Healthcare and for other acute pain and trauma surgery providers.

The aim of this study involves pain management for patients with acute traumatic rib fractures and therefore must involve human subjects.

ELIGIBILITY:
Inclusion Criteria:

- All adult patients admitted to Stanford Health Care with two or more acute traumatic rib fractures.

Exclusion Criteria:

* Hemodynamically instability,
* Mechanical ventilation,
* Polytrauma (defined as bone or organ injury outside the thorax),
* Pregnancy,
* Incarceration
* Local anesthetic allergy or contraindications to lidocaine (Stokes-Adams syndrome, Wolff-Parkinson-White syndrome, or severe degrees of sinoatrial, atrioventricular, or intraventricular block)
* Chronic opioid use.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
OME consumption at 24 hours of treatment. | Up to 24 hours of treatment
  Oral morphine equivalent consumption at 24 hours of treatment

SECONDARY OUTCOMES:
OME at 48 hrs | Up to 48 hours of treatment
  Oral morphine equivalent consumption at 48 hours of treatment
Pain Score | Every 4 hours general pain scores, and baseline, 24 hours, 48 hour, 72 hours for pain scores with cough and inspiration.
  Pain scores at rest and with cough and deep inspiration. Will use Numeric Rating Scale (NRS) of 0-10, where 0 is no pain and 10 is the worst imaginable
Incentive spirometry volumes (volume of 0 - 5000 mL) | Time 0, 24 hours, 48 hour, and 72 hours
  An incentive spirometer is a device that measures how deeply you can inhale. Higher volumes indicate greater ability to inhale.
PIC score | Time 0, 24 hours, 48 hour, and 72 hours.
  PIC score is a composite score comprising pain level, ISV, and cough strength. PIC scores range from 1-10 with one being severe pain, inability to perform incentive spirometry, and absent cough and 10 being controlled pain, an incentive spirometry volume above goal volume(set by respiratory therapist), and strong cough
Length of hospital stay | Up to 10 days
  We will record the number of days stayed at the hospital from the day of operation till the day of discharge (from 0-10, or 10+)
Inflammatory biomarkers | Time 0, 24 hours, and 48 hour
  Will be looking at proinflammatory markers (IL6, IL8, IL-1β, TNF-α) and f anti-inflammatory markers (IL10)
Rates of pulmonary complications | Will be assessed up to 72 hours
  We will look at the occurrence of complications such as ARDS, pneumonia, aspiration, empyema, including need for positive pressure ventilation, pneumonia, aspiration, supplemental oxygen

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Health Care, Stanford, California, United States

REFERENCES:
- [Background] Hollmann MW, Durieux ME. Local anesthetics and the inflammatory response: a new therapeutic indication? Anesthesiology. 2000 Sep;93(3):858-75. doi: 10.1097/00000542-200009000-00038. No abstract available. PMID 10969322
- See also: Aggarwal A. A Role for Peripheral Intravenous Lidocaine Infusion for Rib Fracture Pain Management. Poster presented at: ASRA 16th Annual Pain Medicine Meeting of the Society of Regional Anesthesia and Pain Medicine; Nov 16-18, 2017; Lake Buena Vista, FL. — http://epostersonline.com/ASRAFALL17/node/108